CLINICAL TRIAL: NCT02331732
Title: Virtually Observed Treatment (VOT) for Tuberculosis Patients in Moldova
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Behavioural Insights Team (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 201405*
Record Dates: First submitted 2014-12-13; First posted 2015-01-06 (Estimated); Last update posted 2015-09-25 (Estimated); Status verified 2015-09

CONDITIONS: Tuberculosis
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Active Comparator): Patients receive DOT as normal - involves patient going to polyclinic to be observed taking treatment every day
  Interventions: Other: Directly Observed Treatment
- Treatment (Experimental): Patients receive VOT - involves patient sending a video of themselves taking their treatment over M-health app which will be reviewed remotely by observers
  Interventions: Behavioral: Virtually Observed Treatment

INTERVENTIONS:
Behavioral: Virtually Observed Treatment
  Arms: Treatment
Other: Directly Observed Treatment
  Arms: Control

SUMMARY:
This trial aims to increase the wellbeing of tuberculosis patients and their adherence to medication in Chisinau, The Republic of Moldova. The design is an individually randomised controlled trial (RCT) and will involve 400 TB patients during their 'continuation phase' of treatment. The trial will have two arms; 200 patients will form the control group and receive the standard provision of Directly Observed Treatment (DOT) and 200 will receive Virtually Observed Treatment (VOT).

VOT differs from DOT in that the daily observation of patients taking their medication will be observed via internet video messages rather than in-person. Based on a small sample of patient interviews we think that for some patients DOT may be a hindrance rather than a help. VOT allows patients to take their treatment in the comfort of their home and means they don't have to travel to their polyclinic every day.

There will be a central VOT observation centre where VOT observers will view and respond to video messages sent in by patients in the VOT arm. The messages will be sent via an M-Health app. The VOT observers will also respond to the patients by sending feedback to the patients. The trial duration will depend on the recruitment rate of eligible patients but is expected to take 16 months.

ELIGIBILITY:
Inclusion Criteria:

1. Consent to being part of the trial
2. Live in Chisinau and no plans to move away from Chisinau during the four months
3. Aged 18 or over
4. At least four months of care remaining

Exclusion Criteria:

1. Having MDR-TB
2. Homeless
3. Is not homeless
4. Suffer from alcoholism or drug misuse
5. In prison
6. Has a treatment regimen with injections

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2015-10; Primary Completion 2017-02 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Adherence to medication | 2 weeks
  Number of days per two week period that each patient fails to adhere to treatment, continuous. Panel data collected from TB-01 record sheets for duration of patient continuation phase of treatment - on average 5 months

SECONDARY OUTCOMES:
Adherence 80% | 2 weeks
  Proportion of patients having more than 80% of scheduled medication sessions per two week period (binary). Panel data collected for duration of patient continuation phase of treatment - on average 5 months
Patient wellbeing | Collected at 4 months
  Self reported using a short form version (5 questions) of the WEMWBS questionnaire for measuring mental wellbeing was developed by researchers at Warwick and Edinburgh Universities
Patient satisfaction | Collected at 4 months
  Binary variable equal to 1 if a patient gives a positive response about their treatment on a likert scale (questionnaire, self-reported)
Travel and time cost of treatment borne by patient, self reported. | Collected at 4 months
  Total travel time and cost over 4 months (derived from questionnaire, self-reported)
Employment, self reported | Collected at 4 months
  Binary variable equal to 1 if patient currently does any work for pay or profit (questionnaire, self-reported)
Treatment success | Collected at 4 months
  Binary variable equal to 1 if treatment recorded a success on TB-01 patient record at 4 months
Body mass index (BMI) | Collected at 4 months
  Body mass index (BMI), measured at 4 months
Side effects reported during treatment | Collected at 4 months
  Binary variable equal to 1 if patient reported any side effects during treatment (questionnaire, self-reported)

REFERENCES:
- [Derived] Ravenscroft L, Kettle S, Persian R, Ruda S, Severin L, Doltu S, Schenck B, Loewenstein G. Video-observed therapy and medication adherence for tuberculosis patients: randomised controlled trial in Moldova. Eur Respir J. 2020 Aug 6;56(2):2000493. doi: 10.1183/13993003.00493-2020. Print 2020 Aug. PMID 32381495